CLINICAL TRIAL: NCT06238843
Title: A Multicenter, Randomized, Open-label, Phase 3 Study of IBI343 Monotherapy Versus Treatment of Investigator's Choice in Subjects With Previously Treated, Claudin (CLDN) 18.2-positive, HER2-negative, Locally Advanced, Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Multicenter, Phase 3 Study of IBI343 Monotherapy Versus Treatment of Investigator's Choice in Subjects With Previously Treated, Claudin (CLDN) 18.2-positive, HER2-negative, Gastric or Gastroesophageal Junction Adenocarcinoma
Acronym: G-HOPE-001
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI343A301
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Irinotecan; Paclitaxel; Trifluridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: control arm (Active Comparator): There are three drugs ( irinotecan, paclitaxel,or FTD/TPI (only are applicable in US/EU/Japan and other regions where FTD/TPI is approved for GC treatment)) in active contral arm, the subjects will receive the drug based on investigator's choice
  Interventions: Drug: Irinotecan OR Paclitaxel or Trifluridine/tipiracil（ FTD/TPI）
- IBI343 monotherapy (Experimental): IBI343: Subjects in the experimental arm will receive IBI343 6mg/kg intravenous infusion (IV) D1, Q3W in 3-week cycles .
  Interventions: Drug: IBI343

INTERVENTIONS:
Drug: Irinotecan OR Paclitaxel or Trifluridine/tipiracil（ FTD/TPI） — Drugs: Irinotecan Subjects in the control arm will receive irnotecan 150mg/m2 IV D1, D15, Q4W in 4-weeks cycles.
  Drugs: Paclitaxel Subjects in the control arm will receive paclitaxel 80mg/m2 IV D1, D8, D15, Q4W in 4-week cycles, Drugs:FTD/TPI Subjects in the control arm will receive FTD/TPI 35 mg/m2 up to a maximum of 80 mg orally twice a day on Days 1 to 5 and Days 8 to 12, Q4W (applicable in US/EU/Japan and other regions where FTD/TPI is approved for GC treatment).
  Arms: Active Comparator: control arm
Drug: IBI343 — Subjects in the experimental arm will receive IBI343 6mg/kg intravenous infusion (IV) D1, Q3W in 3-week cycles .
  Other Names: Arcotatug Tavatecan
  Arms: IBI343 monotherapy

SUMMARY:
This is a Multicenter, Randomized, Open-label, Phase 3 Study of IBI343 Monotherapy Versus Treatment of Investigator's Choice in Subjects with Previously Treated Claudin (CLDN) 18.2-positive, HER2-negative, Locally Advanced, Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma to compare the progression free survival (PFS) and overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to sign a written Informed Consent Form(ICF) and to comply with protocol-specified visits and related procedures.
2. Has histopathologically confirmed unresectable locally advanced or metastatic adenocarcinoma of the gastric/gastroesophageal junction (G/GEJ AC).
3. Has received and progressed on at least 2 lines of systemic therapy (anti-PD-(L)1 in combination with platinum or fluoropyrimidines, paclitaxel/docetaxel, irinotecan). A prior (neo)adjuvant systemic therapy that ended within 6 months prior to disease relapse is defined as the first line therapy. The subject has ≤ 4 prior lines of systemic therapy.
4. Has histopathologically confirmed CLDN18.2-positive disease.
5. Is a man or woman of 18 years of age or older at the time of signing the ICF.
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.

Exclusion Criteria:

1. Has HER2-positive (defined as immunohistochemistry [IHC] 3+, or IHC 2+ and positive by in situ hybridization) disease.
2. Is currently participating in another interventional clinical study, except when the subject is during survival follow-up of an interventional clinical study.
3. Has a history of treatment with topoisomerase inhibitorbased antibody-drug conjugate(s).
4. Has received the last dose of an anti-cancer therapy (including traditional Chinese medicine indicated for gastric cancer in the package insert, but excluding herbal prescriptions) within 4 weeks or 5 half-lives (whichever is shorter) prior to the first dose of study treatment.
5. Plans to receive other anti-cancer therapy during treatment with the study drug (palliative radiotherapy for symptomatic (e.g., pain) relief that does not affect response assessment is allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
progression free survival(PFS) | within approximately 20 months
  Progression-free survival (PFS) is defined as the time from random assignment in the trial to disease progression or death from any cause.
overall survival(OS) | within approximately 26 months
  Overall survival (OS) is defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | within approximately 20 months
  ORR is defined as the proportion of subjects in the analysis population who achieve confirmed objective response (CR or PR) as assessed by the IRRC per RECIST v1.1.
disease control rate (DCR) | within approximately 20 months
  DCR is defined as the proportion of subjects in the analysis population who achieve disease control (CR, PR, or SD) as determined by the IRRC per RECIST v1.1 criteria.
duration of response (DoR) | within approximately 20 months
  DoR is defined as the time from the first CR or PR to disease progression or death from any cause, whichever occurs first for subjects with ORR as assessed by IRRC per RECIST v1.1 criteria.
time to response (TTR) | within approximately 20 months
  TTR is defined as the time from randomization to the first CR or PR for subjects with ORR as assessed by IRRC per RECIST v1.1 criteria.
area under the curve (AUC) | within approximately 20 months
  Area under the curve (AUC) is defined as the area under the plasma concentration versus time curve.
maximum concentration (Cmax) | within approximately 20 months
  Cmax is the highest concentration of a drug in the blood after the drug has been administered and before the administration of a second dose.
time to maximum concentration(Tmax) | within approximately 20 months
  The time it takes for a drug to reach the maximum concentration (Cmax) after administration of the drug
trough concentration (Ctrough) | within approximately 20 months
  Ctrough is the lowest concentration of a drug in the blood after the drug has been administered and before the administration of a second dose.
clearance (CL) | within approximately 20 months
  The clearance is defined as the plasma volume in the vascular compartment that is cleared of drug per unit of time.
volume of distribution (V) | within approximately 20 months
  Volume of distribution (Vd) is defined as the arrangement or rate of incidence of a drug in the body in relation to the measured plasma concentration.
Incidence of anti-drug antibody (ADA) | within approximately 20 months
  Incidence of anti-drug antibody (ADA) is defined as the sum of both treatmentinduced (post-baseline ADA-positive only) and treatment-boosted ADA.
neutralizing antibody (NAb) | within approximately 20 months
  Neutralizing antibodies (NAb) are a subset of binding ADA that bind to the drug and inhibit its pharmacological function by preventing target binding.

CONTACTS AND LOCATIONS:
Locations (22):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China
- Japan (21):
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Gunma Prefectural Cancer Center, Ota-Shi, Gunma
  - Kure Medical Center And Chugoku Cancer Center, Kure, Hirosima [Hiroshima]
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Hukuoka [Fukuoka]
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kochi Health Sciences Center, Kochi, Koti [Kochi]
  - Kindai University Hospital, Osakasayama-Shi, Osaka
  - The University of Osaka Hospital, Suita-shi, Osaka
  - Saitama Medical University - International Medical Center, Hidaka-Shi, Saitama
  - Saitama Prefectural Cancer Center, Kitaadachi-Gun, Saitama
  - Chiba Cancer Center, Chiba, Tiba [Chiba]
  - University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - Tokyo Metropolitan Komagome Hospital, Bunkyō-Ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto, Tokyo
  - Gifu University Hospital, Gifu
  - Osaka Prefectural Hospital Organization - Osaka International Cancer Institute, Osaka

IPD SHARING:
Plan to Share IPD: No